CLINICAL TRIAL: NCT02945423
Title: Improving the Understanding of Catatonia in Autism
Acronym: A-CAT
Status: Withdrawn | Type: Observational
Why Stopped: funding issues
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Neera Ghaziuddin, Associate Professor, University of Michigan
Other Study IDs: HUM00113776
Record Dates: First submitted 2016-10-20; First posted 2016-10-26 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Autistic Disorder; Catatonia
MeSH Terms: conditions — Autistic Disorder; Catatonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA: one 8ml vial of blood will be drawn and stored for future DNA analysis. DNA will be stored as part of the Heinz C. Prechter Genetics Repository.Once the DNA is extracted and genotyped, researchers will sequence the genetic information for specific variants. All samples and data will be de-identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Catatonia is a neuropsychiatric syndrome which is frequently missed or misdiagnosed among psychiatric patients. The current project is a systematic examination of catatonia which will characterize the phenotype and identify biological correlates that play a central role in the pathophysiology and effective pharmacological treatment of this condition.

DETAILED DESCRIPTION:
The specific aims of the study are to:

1. Identify and phenotype participants ranging in age from 10-30 years old who are already diagnosed with catatonia.
2. Review laboratory investigations already complete and further conduct any laboratory tests which were not previously completed, to exclude a general medical etiology of catatonia.
3. Obtain skin biopsy for fibroblast from participant to reprogram somatic cells to iPSC (induced pluripotent cell lines) which will be differentiated to cortical neurons for in vitro pharmacological studies against the target tissue.

Up to 30 patients will be consented. Eligibility will be determined through UM medical record screening. When a potential participant is identified, the study team will reach out to the treating clinician to make contact with participant about research interest. Informed consent will be obtained prior to initiation of any study-related procedures. Consent may be emailed at request of potential participants or their representative in advance of a scheduled research appointment for their review. Additionally, informed consent will take place in person both verbally and in writing, with adequate time for participants to ask questions.

Following informed consent, a comprehensive psychiatric interview will be completed to identify overall psychiatric diagnoses and symptoms of catatonia. Based on this evaluation, a decision will be made whether or not the individual is testable or untestable for neurocognitive assessments.

A physical exam will be performed which will include weight, height, waist and head circumference, as well as vital signs that include blood pressure and pulse rate.

Electronic medical record (EMR) will be reviewed to identify any comorbid medical condition, lab results and medications received including the response to each agent. The medical disorders (current or past) may include infective 26 27,28, metabolic/ endocrine 29, autoimmune 30, toxic/ drug related 31 and seizure disorders.

Neuropsychological testing (NP): Standardized, well-validated tests will be used to assess emotional, behavioral and neuropsychological functioning where possible. Clinician completed ratings of autism symptoms will be completed, as well as parental rating scales for autism, general behavioral issues, and quality of life. In addition, each participant will undergo brief face-to face evaluations when catatonic symptoms do not preclude testing covering the domains of intellectual functioning, academic achievement, receptive language, executive functioning, and motor skills. These domains are typically included in neuropsychological testing protocols, are brief, and place minimal demands on participants.

Laboratory tests: Laboratory work up required for the purpose of this study will include CBC, CMP, free T4, TSH, thyroid antibodies, ANA, ASO, CRP, urine toxicology, urine or serum organic acids, Cu and ceruloplasmin, anti-NMDAR receptor antibodies, CMA (chromosomal microarray), fragile X, and EEG. If labs have been performed and are in the participant's medical record, they may be used as part of this study and not re-requested based upon physician judgment.

DNA: one 8ml vial of blood will be drawn and stored for future DNA analysis. DNA will be stored as part of the Heinz C. Prechter Genetics Repository.

Skin biopsy: a skin biopsy will be obtained from a subset of participants who meet inclusion and exclusion criteria.

Assessment: Standardized interviews and questionnaires will be completed by the participant or their representative.

Reliability: will be established between the interviewers, at the level of the interview and by best estimate diagnosis. All available sources of clinical information, including medical records, informant data, the ADOS and the ADI-R, will be independently reviewed by a non-interviewing psychiatrist or psychologist. Reviewers' "best-estimate" diagnoses will be established at regular investigator meetings. If all are in agreement, the consensus diagnosis is confirmed.

Quality Assurance: The PI and co-investigators will review all interviews to check for completeness and accuracy. Interviewers will be given feedback and subjects will be re-contacted as needed to correct problems or complete questions. This will reduce errors and missing data.

ELIGIBILITY:
Inclusion Criteria:

1. Age range = 10 to 30 years.
2. Already diagnosed with Catatonia during 2005 to 2015.
3. Inclusive of current symptoms or have had symptoms in past (symptom

Exclusion Criteria:

1. Onset of catatonia is clearly secondary to general medical condition

-

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be determined through University of Michigan medical record screening. Participants will be both male and female, between the ages of 10-30 years old (inclusive) and will have a previous diagnosis of catatonia, not secondary to a medical condition.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Psychiatric, cognitive and biological identification of catatonia in psychiatric illness | Three months
  Psychiatric, medical, neuropsychological and biological testing will be completed in approximately 30 subjects and analyzed and reviewed by PI and Co-PIs to determine parameters of catatonia diagnosis in psychiatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: Neera Ghaziuddin, M.D., Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: Undecided